CLINICAL TRIAL: NCT01511627
Title: A Randomized Controlled Trial Comparing Postoperative Pain Following Total Abdominal Hysterectomy With General Anesthetic vs. Combined General and Spinal Anesthetic
Brief Title: Randomized Controlled Trial Comparing Postoperative Pain Following TAH With GA vs. Combined GA + SAB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research question was answered by Acta Anaesthesiol Scand 2012; 56: 102-109.
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jacelyn Larson, Faculty, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT GA + SAB for TAH
Record Dates: First submitted 2012-01-09; First posted 2012-01-18 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Hysterectomy
MeSH Terms: interventions — Anesthesia, General; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Anesthesia (Active Comparator)
  Interventions: Drug: General Anesthesia (control group)
- General Anesthesia + Spinal Anesthesia (Experimental)
  Interventions: Drug: General Anesthesia + Spinal anesthesia combined

INTERVENTIONS:
Drug: General Anesthesia + Spinal anesthesia combined — All patients will receive a preoperative multimodal analgesic regime:
  * Tylenol® 975mg per os
  * Naproxen® 500 mg per os
  Patients will receive a spinal anesthetic with:
  * Bupivacaine 0.5% 10 mg
  * Fentanyl 10ug
  * Epidural Morphine 150ug
  After the spinal, a general anesthetic will be induced using:
  * Midazolam 1 - 2 mg intravenously
  * Fentanyl 1 - 2 ug/kg intravenously
  * Propofol 1-3 mg/kg intravenously
  * Rocuronium 0.3 - 0.9mg/kg intravenously
  * followed by endotracheal intubation. Maintenance of anesthesia with sevoflurane, oxygen and air.
  * Intraoperative Morphine 0 - 0.3mg/kg or Fentanyl 0 - 7.5ug/kg to maintain MAP and heart rate within 20% of baseline.
  * Phenylephrine and Ephedrine can be used to support blood pressure and heart rate within 20% of baseline.
  * Dexamethasone 4mg and Ondansetron 4mg intravenously
  * Neostigmine 3mg and Glycopyrrolate 0.6mg intravenously Patients will receive a Morphine PCA to be initiated in the Post Anesthetic Care Unit (PACU).
  Arms: General Anesthesia + Spinal Anesthesia
Drug: General Anesthesia (control group) — All patients will receive a preoperative multimodal analgesic regime:
  * Tylenol® 975mg per os
  * Naproxen® 500 mg per os
  Group I (General anesthetic) patients will receive a general anesthetic :
  * Midazolam 1 - 2 mg intravenously
  * Fentanyl 1 - 2 ug/kg intravenously
  * Propofol 1-3 mg/kg intravenously
  * Rocuronium 0.3 - 0.9mg/kg intravenously
  * followed by endotracheal intubation. Maintenance of anesthesia with sevoflurane, oxygen and air.
  * Intraoperative Morphine 0 - 0.3mg/kg or Fentanyl 0 - 7.5ug/kg. to maintain MAP and heart rate within 20% of baseline.
  * Phenylephrine and Ephedrine can be used to support blood pressure and heart rate within 20% of baseline.
  * Dexamethasone 4mg and Ondansetron 4mg intravenously
  * Neostigmine 3mg and Glycopyrrolate 0.6mg intravenously
  Patients will receive a Morphine PCA as per protocol that will be initiated in the Post Anesthetic Care Unit (PACU).
  Arms: General Anesthesia

SUMMARY:
The investigators hypothesize that a spinal anesthetic administered prior to the induction of general anesthesia will result in reduced need for pain medication and reduced postoperative pain, as well as reduced hospital stay following a total abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists' (ASA) I and II patients undergoing elective Total Abdominal Hysterectomy at the Saskatoon City Hospital
* Lower transverse abdominal incision

Exclusion Criteria:

* BMI > 40
* The TAH is treatment for cancer
* A history of regular opioid use
* Any medical condition that would make a spinal inadvisable,
* An allergy or medical condition that would make it inadvisable to receive the drugs used in this study (eg. Peptic ulcer disease), or
* If you will also be having a salpingo-oophorectomy).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 1 day
  The primary outcome will be total opioid use per day, as recorded by the PCA pump and transcribed by the nursing staff in the PACU and on the post-operative ward.
Total Morphine consumption | Post-operative day 1
  The primary outcome will be total opioid use per day, as recorded by the PCA pump and transcribed by the nursing staff in the PACU and on the post-operative ward.
Total Morphine consumption | Post-operative day 2
  The primary outcome will be total opioid use per day, as recorded by the PCA pump and transcribed by the nursing staff in the PACU and on the post-operative ward.

SECONDARY OUTCOMES:
Pain score on the VAS | In the PACU: within the first 5 minutes
Pain score on the VAS | In the PACU: after 30 minutes
Pain score on the VAS | In the PACU: after 60 minutes.
Pain score on the VAS | Upon arrival on the post-operative ward
Pain score on the VAS | On the post-operative ward: after 1 hour
Pain score on the VAS | On the post-operative ward: after 4 hours
Pain score on the VAS | On post-operative day 1 at 02:00
Pain score on the VAS | On post-operative days 1 at 06:00
Pain score on the VAS | On post-operative days 1 at 10:00
Pain score on the VAS | On post-operative days 1 at 14:00
Pain score on the VAS | On post-operative days 1 at 18:00
Pain score on the VAS | On post-operative days 1 at 22:00
Pain score on the VAS | On post-operative day 2 at 02:00
Pain score on the VAS | On post-operative day 2 at 06:00
Pain score on the VAS | On post-operative day 2 at 10:00
Pain score on the VAS | On post-operative day 2 at 14:00
Pain score on the VAS | On post-operative day 2 at 18:00
Pain score on the VAS | On post-operative day 2 at 22:00

CONTACTS AND LOCATIONS:
Overall Officials: Jacelyn Larson, MD, FRCPC, Principal Investigator — University of Saskatchewan
Locations (1):
- Saskatoon City Hospital, Saskatoon, Saskatchewan, Canada